CLINICAL TRIAL: NCT01816620
Title: An Open-label Phase II Study to Determine the Efficacy and Safety of Lenalidomide Plus Dexamethasone (LDex) in Patients With Newly Diagnosed POEMS Syndrome
Brief Title: Study to Evaluate Lenalidomide Plus Dexamethasone in Patients With Newly Diagnosed POEMS Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Jian Li, Associate professor of Hematology Department, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: POEMS-01
Record Dates: First submitted 2013-03-14; First posted 2013-03-22 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: POEMS Syndrome
Keywords: POEMS Syndrome; lenalidomide; newly diagnosed; plasma cell disorder; Dexamethasone
MeSH Terms: conditions — POEMS Syndrome; Neoplasms, Plasma Cell | interventions — Lenalidomide; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lenalidomide, dexamethasone (Experimental): Lenalidomide 10mg qd d1-21 & dexamethasone 40mg qw d1,8,15,22
  Interventions: Drug: Lenalidomide, Dexamethasone

INTERVENTIONS:
Drug: Lenalidomide, Dexamethasone — 12 cycles of lenalidomide and dexamethasone, each cycle lasts 28 days. For patients with Ccr equal to or higher than 30ml/min, oral lenalidomide 10mg once daily for days 1-21 out of a 28 cycle.
  For patients with Ccr lower than 30ml/min, oral lenalidomide 10mg once every other day for days 1-21 out of a 28 cycle.
  All the patients take Dexamethasone orally 40mg once weekly for day 1,8,15,22 out of a 28 cycle.
  Other Names: Revlimid

SUMMARY:
The purpose of this prospective study is to determine the efficacy and safety of lenalidomide plus dexamethasone in patients with newly diagnosed POEMS syndrome.

DETAILED DESCRIPTION:
The investigators propose to use the adverse effects as well as the need for dose reduction as a criterion to judge tolerability of treatment.

The primary endpoint would be hematological response rate according to international myeloma working group (IMWG) response criteria for amyloidosis and neurological response rate defined by overall neuropathy limitation scale (ONLS) score.

This study expects to enroll approximately 41 subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must understand and voluntarily sign an informed consent form.
2. Older than 18 years old at the time of signing consent.
3. Meet the diagnostic criteria of POEM syndrome.
4. Must be cytotoxic treatment naive. However, previous or existing corticosteroid (prednisone or dexamethasone) or intravenous immunoglobin (IVIG) therapy is allowed.
5. Women of childbearing potential must understand that the study medication could have a potential teratogenic risk. They should undergo complete contraception during the study period.
6. Male subjects must agree to use condoms throughout study drug therapy.

Exclusion Criteria:

1. Any serious medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from signing the informed consent form.
2. Pregnant or lactating females.
3. Any of the following laboratory abnormalities:

   Absolute neutrophil count(ANC) of<1.0×10E9 cell/L. Platelet count<50×10E9 cell/L. Renal failure requiring dialysis. Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3 times of the normal upper limit.
4. Prior history of malignancies, but not including basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, and T1a or T1b prostate cancer.
5. Known hypersensitivity or prior history of uncontrollable side effects to dexamethasone therapy.
6. Prior use of cytotoxic drugs.
7. Subjects who are unable or unwilling to undergo antithrombotic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2015-10 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Hematological response rate | last day of the LDx treatment regimen (up to 9 months)
Neurological response rate defined by ONLS score | last day of the LDx treatment regimen (up to 9 months)

SECONDARY OUTCOMES:
response rate of critical organs | every month during the first 3 months calculated from the day study started, then every 3 months in the next 9 months
Response rate of serum vascular endothelial growth factor (VEGF) level | every month during the first 3 months calculated from the day study started, then every 3 months in the next 9 months
Time to initial neurological response | every month during the first 3 months calculated from the day study started, then every 3 months in the next 9 months
Overall survival | From date of first diagnosis until the date of death from any cause, otherwise patients will be censored in June, 2018 (up to 5 years)
Relapse free survival | From date of first diagnosis until the date of first documented relapse or date of death from any cause, whichever came first, otherwise patients will be censored in June, 2018 (up to 5 years)
adverse events | throughout the treatment and until 30 days after the administration of the last dose of a study drug
time to the best neurological response | every month during the first 3 months calculated from the day study started, then every 3 months in the next 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Jian Li, M.D., Principal Investigator — Peking Union Medical College Hospital; Dao-bin Zhou, MD, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao Y, Zhang S, Yang L, Li J, Liu Y, Wang T. Skin Responses in Newly Diagnosed Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal Gammopathy, and Skin Changes (POEMS) Syndrome After Therapy With Low-Dose Lenalidomide Plus Dexamethasone. Front Immunol. 2021 May 6;12:681360. doi: 10.3389/fimmu.2021.681360. eCollection 2021. PMID 34025681
- [Derived] Liu LS, Zhang X, Zhao H, Gao XM, Zhou DB, Dai RP, Li J. Reliability of optic disc edema area in estimating the severity of papilledema in patients with POEMS syndrome. Orphanet J Rare Dis. 2020 May 19;15(1):116. doi: 10.1186/s13023-020-01392-x. PMID 32429967
- [Derived] Li J, Huang XF, Cai QQ, Wang C, Cai H, Zhao H, Zhang L, Cao XX, Gale RP, Zhou DB. A prospective phase II study of low dose lenalidomide plus dexamethasone in patients with newly diagnosed polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes (POEMS) syndrome. Am J Hematol. 2018 Jun;93(6):803-809. doi: 10.1002/ajh.25100. Epub 2018 Apr 18. PMID 29603764